CLINICAL TRIAL: NCT00912275
Title: Phase I/II Study of Lapatinib in Combination With Oral Vinorelbine for Metastatic Breast Cancer
Brief Title: Lapatinib in Combination With Oral Vinorelbine for Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200811019M
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib plus Oral Vinorelbine (Experimental): Oral vinorelbine on day 1 and day 8 q3w plus lapatinib 1000mg/day.
  Interventions: Drug: lapatinib plus oral vinorelbine

INTERVENTIONS:
Drug: lapatinib plus oral vinorelbine — Lapatinib -dose level -I, I, II, III 1000mg po daily;dose level IV:1250mg po daily; Oral vinorelbine at the dose level reached on days 1, and 8 of a 21 days cycle. Dose level -I:30mg/m2,I:40mg/m2,II:50mg/m2,III:60mg/m2,IV:60mg/m2,V:80mg/m2
  Other Names: Tykerb, Navelbine

SUMMARY:
Phase I part: to determine the recommended dose, and observe the preliminary response and safety profile of the combination of oral lapatinib with vinorelbine in patients with ErbB2 positive metastatic breast cancer.

Phase II part: to determine the progression free survival, response rate, and to evaluate the safety profile of the combination of oral lapatinib with vinorelbine in patients with ErbB2 positive metastatic breast cancer.

Phase I part has been completed. Phase II part is underway.

DETAILED DESCRIPTION:
This is a phase I/II clinical trial. In phase I part, the primary objective is To determine the recommended dose of the combination of lapatinib with oral vinorelbine in patients with ErbB2 positive metastatic breast cancer. In phase II part, the primary objective is progression free survival of the combination of lapatinib with oral vinorelbine as first line chemotherapy in patients with ErbB2 positive metastatic breast cancer. The secondary objectives are safety profile and the response rate

Lapatinib, an oral inhibitor of EGFR and HER2, have been shown to be an effective treatment in HER2/neu overexpressing metastatic breast cancer patient who refractory herceptin, taxane, and anthracycline treatment. In pre-clinical studies, the highest synergism between anti-Her2 treatment (trastuzumab) and cytotoxics was seen with the platinum compounds and with vinorelbine. The oral vinorelbine has similar efficacy to that of the injection formulation and has demonstrated generally favorable tolerability. We are interested in lapatinib plus oral vinorelbine as 1st line treatment in Her2+ MBC, to which we believe this convenience treatment offer a good response rate with satisfactory life quality.

For phase I part, we plan to use the standard phase I 3-patient cohort (''3 + 3'') design. Up to 18 patients may be enrolled. For phase II part, the expected progression-free survival of the protocol treatment in first line treatment of ErbB2 positive metastatic breast cancer is more than 6 months. With type 1 and type 2 errors of 0.05 and 0.1, respectively, this design calls for 29 patients at the first stage. If 20 or more progression disease is observed after 6 months of treatment, then the study will be terminated. Otherwise, additional 25 patients will be entered at the second stage. The treatment will be rejected if a total of 37 or more progression disease are observed out of 54 patients after 6 months of treatment. With the estimated dropout rate of 10%, 32 patients will be accrued in the first stage and 28 in the second stage.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the breast which is now metastatic.
2. Documented ErbB2 over expression or amplified disease in the invasive component of the primary or metastatic lesion as defined by:

   * 3+ over expression by IHC or
   * ErbB2 gene amplification by FISH/CISH (> 6 ErbB2 gene copies per nucleus, or a FISH ratio (ErbB2 gene copies to chromosome 17 signals) of > than 2.2;
3. In phase II part, patients must be chemo-naïve in metastatic setting. In phase I part, patient may have received prior chemotherapy including vinorelbine in metastatic setting. However, patient must be informed and well understand that in current standard of treatment, suggested first line treatments for erbB-2 positive, visceral organ metastatic breast cancer are combination of chemotherapy with herceptin.
4. In phase II part, patient must not have exposed to ant-erbB2 targeted therapy treatment in metastatic setting. Herceptin treatment in the neoadjuvant or adjuvant setting is permitted provide that at least 12 months has elapsed since the last dose of herceptin therapy. In phase I part, patient may have received prior anti-erbB-2 targeted treatment in metastatic setting.
5. Prior treatment with endocrine therapy in the adjuvant or metastatic setting permitted provided that therapy has been discontinued.
6. Prior treatments with radiation therapy for palliative management of metastatic disease permitted provided that at least 2 weeks have elapsed since the last fraction of radiation therapy, disease progression has been documented and all treatment related adverse events are < grade 1 at the time of registration.
7. Patients must have evidence of metastatic disease, but measurable disease is not mandatory. To be considered evaluable for the overall response rate (complete and partial response), patients must have at least one measurable lesion as follows:

   * X-ray, physical exam >= 20 mm
   * Conventional CT scan, MRI >= 20 mm
   * Spiral CT scan >= 10 mm
8. Age > 20 years.
9. Life expectancy > 3 months.
10. ECOG PS 0-2.
11. Patients must have normal organ and marrow function measured within 14 days prior to randomization as defined below:

    * Hemoglobin>10.0;
    * Absolute neutrophil count > 1,500/uL;
    * Platelets >75,000/uL;
    * Total bilirubin <= 1.5 X upper normal limit;
    * AST(SGOT)/ALT(SGPT) <= 2.5 X upper normal limit;
    * Creatinin <= 1.5 X upper normal limit;
    * Patient must have cardiac ejection fraction > 50% and within the institutional range of normal as demonstrated by MUGA scan/echocardiogram within 4 weeks of registration.
12. CT or MRI within 4 weeks prior to randomization.
13. Women of childbearing potential must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to registration.
14. Patient consent must be obtained.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
3. Prior therapy with lapatinib.
4. CNS metastases.
5. Ongoing anticancer treatment.
6. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious non-healing wound/ulcer/bone fracture, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11-24 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
To determine the recommended dose of the combination of oral lapatinib with vinorelbine (phase I part), and progression free survival (phase II part) | phase I part: 4 months, phase II part: 1 and half years

SECONDARY OUTCOMES:
response rate, safety profile | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, M.D.,Ph.D, Principal Investigator — Department of Oncology,National Taiwan University Hospital
Locations (1):
- Department of Oncology,National Taiwan University Hospital, Taipei, Taiwan